CLINICAL TRIAL: NCT05932433
Title: Effectiveness of Therapeutic Exercise on the Gut Microbiome in Chronic Widespread Pain Patients.
Acronym: MiBioPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, María Elena González Álvarez, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1601202303523
Record Dates: First submitted 2023-06-22; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Arthritis; Fibromyalgia; Arthritis Rheumatoid; Artrosis of the Knee; Chronic Pain; Central Sensitisation; Gut Microbiota; Exercise Therapy
MeSH Terms: conditions — Arthritis; Fibromyalgia; Arthritis, Rheumatoid; Chronic Pain | interventions — Exercise; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercise during 6 weeks, twice a week.
  Interventions: Behavioral: Exercise
- Control (No Intervention): There is no intervention

INTERVENTIONS:
Behavioral: Exercise — Each session (45 minutes aprox) is made by: mobility, endurance and final exercise to rest. The sesion is going to perform twice a week during 6 weeks.
  Other Names: Therapeutic exercise; physical activity
  Arms: Exercise

SUMMARY:
This study aims to evaluate the effect of therapeutic exercise on the gut microbiome in chronic widespread pain patients. Our investigation purpose is to improve the quality of life of participants, reduce their disability and optimize their functionality.

The intervention will last 6 weeks, with 2 face-to-face therapeutic exercise sessions guided by a professional and a 6-week post-intervention follow-up.

The participation will require:

1. Attend the 12 therapeutic exercise sessions
2. Attend the 3 evaluations: at the beginning (A0), post intervention (A1) and +6 weeks after finishing the exercise program (A3).

The items to be evaluated will be the following:

1. The Ronald Morris Disability Questionnaire (RMDQ)
2. Anxiety (State-Trait Anxiety Inventory (STAI))
3. Depression: Beck Depression Inventory (BDI)
4. Quality of Life: SF-12
5. Pain: numerical scale (0-100) and The Brief Pain Inventory (BPI)
6. Sensory tests: heat pain threshold (HPT), pressure pain threshold (PPT) and pain modulation (CPM)
7. Perform a pre blood test on interleukins IL-18 and IL-1β

This study involves the processing of personal data, so the researchers will guarantee confidentiality in their treatment at all times, complying with the personal data protection regulations, in particular, European Regulation 679/2016. , of April 27, general data protection, as well as Organic Law 3/2018, of December 5, Protection of Personal Data and Guarantee of Digital Rights.

In order to maintain your privacy and anonymity during the research, only one person on the research team will know how names were assigned to a participation number.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years old
* Must be diagnosed with: osteoarthritis, osteoarthritis, Sudeck or fibromyalgia.

Exclusion Criteria:

* Suffering or having suffered from cancer, psychiatric disorders, or another ongoing major illness (irritable bowel syndrome, hepatitis, Lyme disease or diabetes).
* Patients will be excluded if they have more than 6 points on the Beck Depression Inventory, more than 30 points on the "State Trait Anxiety Inventory" or suffer from dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Quantitative Sensory Test (QST), and | From enrollment to the end of the intervention at 6 weeks
  Conditioned Pain Modulation (CPM) and pain threshold will be assesed as measured of QST.
Psychological and PainTest | From enrollment to the end of the intervention at 6 weeks
  Furthermore,Beck Depression Inventory and State-Trait Anxiety Inventory (STAI) will be perform as a psychological test. The Brief Pain Inventory (BPI) and a numerical rate scale will be perform as a pain tests.
Descriptive parameters | From enrollment to the end of the intervention at 6 weeks
  Descriptive parameters of the sample will be explain in a table

SECONDARY OUTCOMES:
Interleukin analysis | From enrollment to the end of the intervention at 6 weeks
  Interleukin-18 and interleukin-1β analysis will be perform in tha baseline in control group and at the end of the intervention in the experimental (exercise) group

CONTACTS AND LOCATIONS:
Overall Officials: Jorge H Jorge Hugo Villafañe, Dr., Study Director — Responsable científico, Centro "S. Maria ai Colli" - Presidio Ospedaliero "Ausiliatrice", Torino, de la Fondazione Don Carlo Gnocchi Onlus, Italia.
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data and its interpretation are going to be publicated in the Scientific Community through specific and scientific Journals about this topic and Congress.
Supporting Information: Study Protocol, SAP, ICF